CLINICAL TRIAL: NCT06433219
Title: An Open-label, Multicenter, Randomized Phase 2 Study of the ATR Inhibitor Tuvusertib in Combination With the PARP Inhibitor Niraparib or the ATM Inhibitor Lartesertib in Participants With BRCA Mutant and/or Homologous Recombination deﬁciency (HRD)-Positive Epithelial Ovarian Cancer That Progressed on Prior PARP Inhibitor Therapy (DDRiver EOC 302)
Brief Title: Tuvusertib Combined With Niraparib or Lartesertib in Participants With Epithelial Ovarian Cancer (DDRiver EOC 302)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201924_0002; 2024-511202-23-00 (Other: EU trial number)
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
Keywords: Ataxia telangiectasia mutated Rad3-related; Ataxia telangiectasia mutated; Poly-ADP ribose polymerase inhibitor resistance; Homologous recombination deficiency
MeSH Terms: conditions — Ovarian Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A, Arm 1: Tuvusertib with Niraparib (Experimental): In Part A, participants will be randomized to one of 2 arms to receive tuvusertib in combination with either niraparib or lartesertib.
  Interventions: Drug: Tuvusertib (M1774); Drug: Niraparib
- Part A, Arm 2: Tuvusertib with Lartesertib (Experimental): In Part A, participants will be randomized to one of 2 arms to receive tuvusertib in combination with either niraparib or lartesertib.
  Interventions: Drug: Tuvusertib (M1774); Drug: Lartesertib (M4076)
- Part B (dose optimization), dosing regimen 1 :Tuvusertib+Niraparib or Tuvusertib +Lartesertib (Experimental): In Part B, the most favorable combination treatment from Part A will be further explored at 2 different dosing regimens and compared to tuvusertib monotherapy.
  Interventions: Drug: Tuvusertib (M1774); Drug: Niraparib; Drug: Lartesertib (M4076)
- Part B (dose optimization), dosing regimen 2: Tuvusertib + Niraparib or Tuvusertib + Lartesertib (Experimental): In Part B, the most favorable combination treatment from Part A will be further explored at 2 different dosing regimens and compared to tuvusertib monotherapy.
  Interventions: Drug: Tuvusertib (M1774); Drug: Niraparib; Drug: Lartesertib (M4076)
- Part B: Tuvusertib Monotherapy (Experimental): In Part B, the most favorable combination treatment from Part A will be further explored at 2 different dosing regimens and compared to tuvusertib monotherapy.
  Interventions: Drug: Tuvusertib (M1774)

INTERVENTIONS:
Drug: Tuvusertib (M1774) — Tuvusertib will be administered orally.
  Other Names: M1774, VXc-400, VRT-1363004, substance code MSC2584415A
Drug: Niraparib — Niraparib will be administered orally. If selected from Part A, Niraparib will be administered orally in combination with Tuvusertib.
  Other Names: GSK3985771, MK-4827
  Arms: Part A, Arm 1: Tuvusertib with Niraparib; Part B (dose optimization), dosing regimen 1 :Tuvusertib+Niraparib or Tuvusertib +Lartesertib; Part B (dose optimization), dosing regimen 2: Tuvusertib + Niraparib or Tuvusertib + Lartesertib
Drug: Lartesertib (M4076) — Lartesertib will be administered orally. If selected from Part A, Lartesertib will be administered orally in combination with Tuvusertib
  Other Names: M4076, substance code MSC2585823A
  Arms: Part A, Arm 2: Tuvusertib with Lartesertib; Part B (dose optimization), dosing regimen 1 :Tuvusertib+Niraparib or Tuvusertib +Lartesertib; Part B (dose optimization), dosing regimen 2: Tuvusertib + Niraparib or Tuvusertib + Lartesertib

SUMMARY:
The purpose of this study is to measure the effect and safety of treatment with tuvusertib combined with either niraparib or lartesertib in participants with epithelial ovarian cancer and to assess any differences between tuvusertib monotherapy and combination therapy. The participants will previously have progressed while treated with a poly ADP ribose polymerase (PARP) inhibitor. The primary objectives of this study are to assess the effect of the treatment in terms of overall response, i.e. whether the tumor disappears, shrinks, remains unchanged, or gets worse and safety in terms of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed high grade serous or high grade endometrioid ovarian, primary peritoneal, and/or fallopian tube cancer that is recurrent.
* Participants whose tumor carries germline or somatic deleterious or suspected deleterious mutations in the genes BRCA1 (Breast Cancer gene 1) and BRCA2 (Breast Cancer gene 2), and/or tumors with positive HRD status. The presence of any of these mutations and/or the homologous recombination deficiency (HRD) status will be determined according to routinely used local standard of care tests. Results must be available before screening.
* Radiologically confirmed/documented disease progression while on Poly (ADP-ribose) polymerase (PARP) inhibitors therapy in either first or second-line maintenance setting (only 1 line of PARPi maintenance is allowed with or without bevacizumab). Note: Documentation of disease progression must be within 28 days of last PARPi dose taken. Surgical salvage intervention and/or focal ablative therapies are allowed, (further disease progression after these interventions must be documented), AND Clinically benefited from PARPi maintenance prior to documented progression, as defined by at least 6 months of treatment duration with no progressive disease observed, AND either, Progression on first-line maintenance PARPi: Participants are allowed maximum 1 additional line of platinum-based chemotherapy before study entry. (note: treatment-free interval on platinum rechallenge must be >6 months, with documented disease progression prior to study entry).

OR Progression on second-line maintenance PARPi: Participants are not allowed any additional systemic anticancer treatments before study entry (that is PARPi is the last treatment before study entry)

* Intolerant to standard of care treatment options or refused standard of care treatment or the participant's treating physician considers that the lack of standard of care treatment is not detrimental for the participant.
* Measurable disease per RECIST v1.1, as assessed by Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and a life expectancy of at least 6 months.
* Other Protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Primary platinum-refractory disease defined as disease progression during primary platinum-based chemotherapy or platinum-resistant disease defined as disease progression within 6 months of the platinum administration in either the first or second-line setting.
* History of additional malignancy within 3 years before the date of enrollment.
* Known brain metastases, unless clinically stable, that is without evidence of progression by imaging for at least 4 weeks prior to the first dose of study intervention, no evidence of new brain metastases, and on a stable or decreasing dose of ≤ 10 mg of prednisone (or equivalent) or without corticosteroids for at least 14 days prior to study intervention administration.
* Active and/or uncontrolled infection.
* History of known hypersensitivity to the active substances or to any excipients (e.g. polysorbate 80) of the study interventions.
* Organ transplantation, including allogenic stem cell transplant.
* Patients with history of drug-induced severe cutaneous adverse reaction (SCAR; including but not limited to Stevens-Johnson syndrome/toxic epidermal necrolysis [SJS/TEN], or drug reaction with eosinophilia and systemic symptoms [DRESS]), or dose-limiting immune-mediated reactions related to skin.
* Other Protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2028-01-10 (Estimated); Study Completion 2028-01-25 (Estimated)

PRIMARY OUTCOMES:
Part A and Part B: Confirmed Objective Response (OR) According to RECIST v1.1 as Assessed by Investigator | Time from randomization to final assessment or until progressive disease, death, discontinuation criteria, approximately up to 3.5 years
Part A and Part B: Number of Participants With Treatment-Emergent Adverse Events (TEAE), Serious TEAEs and Related TEAEs | Time from randomization to final assessment at end of safety follow-up visit, approximately up to 3.5 years

SECONDARY OUTCOMES:
Part A and Part B: Duration of Response (DoR) According to RECIST 1.1 as Assessed by the Investigator | Time from randomization to final assessment or until progressive disease, death, discontinuation criteria, approximately up to 3.5 years
Part A and Part B: Progression Free Survival (PFS) According to RECIST 1.1 as Assessed by the Investigator | Time from randomization to final assessment or until progressive disease, death, discontinuation criteria, approximately up to 3.5 years
Part B: Overall Survival | Time from date of randomization to death, approximately 3.5 years
  OS is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (84):
- United States (9):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Francisco - UCSF Medical Center, San Francisco, California
  - Centricity Research Cancer Center - DBA CRRI John B. Amos Cancer Center Research, Columbus, Georgia
  - University of Chicago Comprehensive Cancer Center at Silver Cross - Carolyn J. Czerkies Pavilion, Chicago, Illinois
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai PRIME - Mount Sinai - PRIME, New York, New York
  - Next Oncology - Virginia, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown
  - St George Private Hospital, Kogarah
  - Liverpool Hospital - PARENT, Liverpool
- Belgium (2):
  - Cliniques Universitaires Saint-Luc - STL, Brussels
  - UZ Leuven, Leuven
- Denmark (3):
  - Ålborg Universitets Hospital - PARENT, Aalborg
  - Rigshospitalet, Copenhagen
  - Sjaellands Universitetshospital - other, Odense
- France (13):
  - ICO - Site Paul Papin - service d'oncologie medicale, Angers
  - Centre Francois Baclesse - Service d'Oncologie Medicale, Caen
  - Centre Oscar Lambret - service de cancerologie gynecologique, Lille
  - Centre Leon Berard - Service d'Oncologie Medicale, Lyon
  - Groupe Hospitalier Diaconesses - Hôpital De La Croix Saint Simon - service d'oncologie medicale, Paris
  - Hopital Tenon - service d'oncologie medicale, Paris
  - Hôpital Cochin - Hematologie et Oncologie Médicale, Paris
  - Hôpital Européen Georges Pompidou - Hématologie Oncologie, Paris
  - Hôpital Saint Joseph - Paris - Service d'Oncologie-Cancerologie, Paris
  - Centre Hospitalier Lyon Sud - service d'oncologie medicale, Pierre-Bénite
  - Centre de Radiotherapie Clinique Sainte Anne - 300207251, Strasbourg
  - Institut de Cancérologie de Strasbourg Europe - ICANS - Service d'oncologie médicale, Strasbourg
  - Institut Gustave Roussy - Oncologie Médicale, Villejuif
- Germany (9):
  - Charité - Campus Virchow-Klinikum - Klinik fuer Gynaekologie, Berlin
  - Universitaetsklinikum Bonn AoeR - Frauenklinik, Bonn
  - Universitaetsklinikum Carl Gustav Carus TU Dresden - Klinik u. Poliklinik f. Frauenheilkunde, Dresden
  - Kliniken Essen-Mitte - Gynaekologie und Gynaekologische Onkologie, Essen
  - Universitaetsklinikum Leipzig AoeR - Klinik und Poliklinik fuer Frauenheilkunde, Leipzig
  - Universitaetsklinikum Muenster - Parent, Münster
  - Universitätsklinikum Münster - Gynecology, Münster
  - Caritas-Krankenhaus St. Josef - Klinik fuer Chirurgie, Regensburg
  - Universitaetsklinikum Tuebingen - Parent, Tübingen
- Israel (5):
  - Rambam Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Shaare Zedek, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (10):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS - Oncologia Medica, Bologna
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant Orsola - SSD Oncologia Medica Zamagni, Bologna
  - Osp Cannizzaro Catania, Catania
  - Azienda Ospedaliero-Universitaria Renato Dulbecco - Centro Oncologico, Catanzaro
  - IEO Istituto Europeo di Oncologia - Unità Ginecologia Oncologica Medica, Milan
  - Istituto Clinico Humanitas - U.O. di Oncologia Medica ed Ematologia, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale - Gynecology, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS - Radiologia Oncologica, Padua
  - Istituto Nazionale Tumori Regina Elena IRCCS - UOC Oncologia Medica A, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Ostetricia e ginecologia, Rome
- Catharina Ziekenhuis Eindhoven - Parent, Eindhoven, Netherlands
- Poland (6):
  - Centrum Onkologii im. Prof. F. Lukaszczyka w Bydgoszczy - Dept of Chemotherapy, Bydgoszcz
  - Szpitale Pomorskie spó, Gdynia
  - Jagiellonskie Centrum Innowacji Sp. z o.o. - Centrum Bada, Krakow
  - Instytut MSF Sp.z.o.o, Lodz
  - Europejskie Centrum Zdrowia - Oddzial Onkologii, Otwock
  - MICS Centrum Medyczne Torun - Medicovernn, Torun
- Spain (8):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol - Servicio de Oncologia Medica, Badalona
  - Hospital Clinic de Barcelona - Servicio de Oncologia, Barcelona
  - Hospital Universitari Vall d'Hebron - Oncology Dept., Barcelona
  - ICO Girona - Hospital Universitari de Girona Dr Josep Trueta - Servicio de Oncologia Medica, Girona
  - Clinica Universidad de Navarra (MAD) - Oncology Service, Madrid
  - Hospital Universitario 12 de Octubre - Servicio de Oncologia, Madrid
  - Hospital Universitario Ramon y Cajal - Servicio de Oncologia, Madrid
  - Hospital Regional Universitario de Malaga - Oncology Dept, Málaga
- Switzerland (5):
  - Istituto Oncologico della Svizzera Italiana (IOSI)- Ente Ospedaliero Cantonale (EOC) - Ospedale S.Giovann, Bellinzona
  - Kantonsspital Frauenfeld - 150509250, Frauenfeld
  - Kantonsspital Baselland - standort Liestal - Klinik fuer Onkologie, Liestal
  - Kantonsspital St. Gallen - Klinik fuer Med. Onkologie/Haematologie, Sankt Gallen
  - Universitaetsspital Zuerich - Klinik fuer Gynaekologie, Zurich
- United Kingdom (10):
  - Addenbrooke's Hospital - Dept of Oncology, Cambridge
  - Beatson West of Scotland Cancer Centre - Dept of Medical Oncology, Glasgow
  - Royal Surrey County Hospital - Dept of Oncology, Guildford
  - St James's University Hospital - Dept of Oncology, Leeds
  - Guy's Hospital - Dept of Medical Oncology, London
  - Royal Marsden Hospital-London - Dept of Haematology/Oncology Research, London
  - University College London Hospitals - NIHR/Wellcome Trust, London
  - The Christie Hospital - Dept of Oncology, Manchester
  - Mount Vernon Hospital - Dept of Oncology, Northwood
  - Royal Marsden Hospital-Sutton - Dept of Oncology (Surrey), Sutton

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201924_0002
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html